CLINICAL TRIAL: NCT01399281
Title: Pharmacovigilance in Juvenile Idiopathic Arthritis Patients (Pharmachild) Treated With Biologic Agents and/or Methotrexate. A PRINTO/PRES Registry
Brief Title: Pharmacovigilance in Juvenile Idiopathic Arthritis Patients Treated With Biologic Agents and/or Methotrexate
Acronym: PharmaChild
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Giannina Gaslini (Other)
Collaborators: Members of the PRINTO network (PRINTO at www.printo.it) (Unknown)
Responsible Party: Principal Investigator, Dr. Nicola Ruperto, MD, MPH, Istituto Giannina Gaslini
Other Study IDs: EU 260353
Record Dates: First submitted 2011-07-19; First posted 2011-07-21 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: juvenile idiopathic arthritis, biologics, methotrexate
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Biologics alone or methotrexate alone: This group mainly refer to children with polyarticular course JIA treated with methotrexate ± biologics,
- Biologics and MTX: JIA treated with a combination of biologic and MTX (including any other add on therapy e.g. cyclosporine, leflunomide etc). This group mainly refer to children with polyarticular course JIA treated with MTX ± biologics
- NSAIDs and/or steroid injections alone: This group refers to children with mostly oligoarticular persistent course who are usually NOT treated with second line agents and have a more benign course.

SUMMARY:
BACKGROUND: Juvenile idiopathic arthritis (JIA) is the most common chronic paediatric rheumatic disease (PRD) and an important cause of short and long-term disability. Although none of the available drugs for JIA has a curative potential, prognosis has greatly improved as a result of substantial progress in disease management. The therapeutic treatment of children with JIA encompasses the use of NSAIDs and intra-articular steroid injections. In those patients not responding to NSAIDs, methotrexate (MTX) has become the disease modifying anti-rheumatic drug (DMARD) of first choice worldwide. For children not responding to MTX, biologic agents recently have become treatment options.

PATIENTS AND METHODS: 3-10 year observation study related to children with JIA undergoing treatment with MTX or biologic agents with the following objectives:

1. To create a long-term observational registry of a large population of prevalent and incident cases.
2. Use the accumulating data in the registry to conduct (i) a pharmacovigilance/safety study (primary endpoint) and (ii) estimate effectiveness (frequency and magnitude of response, disease activity over time inhibition or slowing of joint erosions and other radiological evidence of disease progression,), and (iii) estimate adherence to the various treatment regimens. Data from the registry will be used to compare safety and effectiveness profiles amongst the patient cohorts.
3. To identify clinical and laboratory predictors of safety, response to therapy, including remission This project has retrospective (first 3 years) and prospective components (up to 10 years) and will be conducted by the participating centres of the more than 50 countries belonging to the Paediatric Rheumatology INternational Trials Organisation (PRINTO certified ISO 9001-2008, www.printo.it), or the Pediatric Rheumatology European Society (PRES at www.pres.org.uk). The main role of these organisations is to provide a scientific basis for current treatments of paediatric rheumatic diseases.

The overall hypothesis to be tested is:

• Biologic agents ± MTX agents are able to maintain an acceptable safety profile in the long term in children with different JIA categories while achieving clinical remission and prevent/stop joint erosion development over time.

The overall aims are to establish the long term safety of biologic agents and MTX, and their relative effectiveness in children with JIA who need treatment with second line agents.

DETAILED DESCRIPTION:
Study Design This is a 3-10 year, international, multicentre, observational, safety and efficacy (response, joint erosion, damage, and treatment adherence) study aimed at collecting prospective safety, tolerability, efficacy, and treatment adherence information on JIA subjects exposed to any biologic agents and MTX, according to local standard of practice.

This is a non-interventional study, where the medicinal products are prescribed as per the investigator's decision. The assignment of the subject to a particular therapeutic strategy is not decided in advance by the study protocol, but falls within current practice and the prescription of the medicine is clearly separated from the decision to include the subject in the study. No additional diagnostic or monitoring procedures shall be applied to the subjects and epidemiological methods will be used for the analysis of collected data.

Duration and treatment will be as per investigator's decision. The nature and frequency of subjects' visits to the investigator's site will be determined only by the investigator, according to his/her judgment on the basis of the clinical evolution of the subject.

The duration of the study is expected to be at least 3 years from initiation of the first site and may be continued beyond if adequate funding is be available.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent by subjects and /or parent or legally acceptable representative;
* JIA (any ILAR category);
* Subjects receiving biologic agents ± MTX, MTX alone, or NSAIDs and/or steroid injections only as per physician discretion.

Exclusion Criteria:

* Contraindications to biologic agents and/or MTX treatment

Ages: 6 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Male and female JIA patients selected among the PRINTO centres as part of the routine standard of care
Sampling Method: Probability Sample
Enrollment: 9000 (Estimated)
Dates: Start 2011-12; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Safety in patients with JIA on biologics/MTX from 3 to 10 years from drug initiation | 3-10 years
  To compare the long term incidence rates of emergent moderate, severe adverse events (AEs) and serious A (SAE) observed in paediatric subjects with JIA. This will include but not be limited to, malignancies, opportunistic infections, autoimmune events, cardiovascular events, central nervous system involvement (e.g. optic neuritis, demyelinating disease), infertility, gastrointestinal bleeding, macrophage activation syndrome (MAS).
Long-term efficacy in patients with JIA on biologics/MTX from 3 to 10 years from drug initiation | 3-10 years
  To assess the long-term efficacy (magnitude of response, prevention or slowing of joint erosion and damage, and treatment adherence) of biologic agents and MTX for the treatment of children and adolescents with different categories of JIA.

SECONDARY OUTCOMES:
Predictors of safety from 3 to 10 years from drug initiation | 3-10 years
  Identify predictors of safety (clinical or experimental, magnitude of response, remission)
Risk factor from 3 to 10 years from drug initiation | 3-10 years
  Assess potential risk factors (e.g. concomitant medications or diseases, medical history etc), which may modify the safety profile of biologic agents and MTX;
Number of children in treatment with biologics from 3 to 10 years from drug initiation | 3-10 years
  To assess the number of children in which a biologic agent is added to the treatment
Wrist joint erosion from 3 to 10 years from drug initiation | 3-10 years
  Evaluate the progression of wrist joint erosion over time and abnormal growth/maturation in JIA subjects presenting a wrist involvement
Assess the reasons for stopping drug treatment from 3 to 10 years from drug initiation | 3-10 years
  • To assess the reasons for stopping drug treatment
Efficacy from 3 to 10 years from drug initiation | 3-10 years
  • To evaluate efficacy in terms, in the different JIA categories, of individual JIA core set variables, and the ACR Paediatric 30, 50, 70, 90, 100 criteria for improvement, and the achievement of clinical remission on and off medication as well as the occurrence of disease flare during biologic agents and MTX treatment course and after drug discontinuation, and the attainment of a status of minimal disease actvity (MDA)

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Ruperto, MD, MPH, Principal Investigator — Istituto G. Gaslini/ PRINTO; PRINTO Member, Study Director — All PRINTO members who will receive ethics committee approval
Locations (1):
- IRCCS G. Gaslini, Genoa, Italy

REFERENCES:
- [Background] Ravelli A, Martini A. Juvenile idiopathic arthritis. Lancet. 2007 Mar 3;369(9563):767-778. doi: 10.1016/S0140-6736(07)60363-8. PMID 17336654
- [Background] Giannini EH, Brewer EJ, Kuzmina N, Shaikov A, Maximov A, Vorontsov I, Fink CW, Newman AJ, Cassidy JT, Zemel LS. Methotrexate in resistant juvenile rheumatoid arthritis. Results of the U.S.A.-U.S.S.R. double-blind, placebo-controlled trial. The Pediatric Rheumatology Collaborative Study Group and The Cooperative Children's Study Group. N Engl J Med. 1992 Apr 16;326(16):1043-9. doi: 10.1056/NEJM199204163261602. PMID 1549149
- [Background] Ruperto N, Murray KJ, Gerloni V, Wulffraat N, de Oliveira SK, Falcini F, Dolezalova P, Alessio M, Burgos-Vargas R, Corona F, Vesely R, Foster H, Davidson J, Zulian F, Asplin L, Baildam E, Consuegra JG, Ozdogan H, Saurenmann R, Joos R, Pistorio A, Woo P, Martini A; Pediatric Rheumatology International Trials Organization. A randomized trial of parenteral methotrexate comparing an intermediate dose with a higher dose in children with juvenile idiopathic arthritis who failed to respond to standard doses of methotrexate. Arthritis Rheum. 2004 Jul;50(7):2191-201. doi: 10.1002/art.20288. PMID 15248217
- [Background] Lovell DJ, Giannini EH, Reiff A, Cawkwell GD, Silverman ED, Nocton JJ, Stein LD, Gedalia A, Ilowite NT, Wallace CA, Whitmore J, Finck BK. Etanercept in children with polyarticular juvenile rheumatoid arthritis. Pediatric Rheumatology Collaborative Study Group. N Engl J Med. 2000 Mar 16;342(11):763-9. doi: 10.1056/NEJM200003163421103. PMID 10717011
- [Background] Ruperto N, Lovell DJ, Cuttica R, Wilkinson N, Woo P, Espada G, Wouters C, Silverman ED, Balogh Z, Henrickson M, Apaz MT, Baildam E, Fasth A, Gerloni V, Lahdenne P, Prieur AM, Ravelli A, Saurenmann RK, Gamir ML, Wulffraat N, Marodi L, Petty RE, Joos R, Zulian F, McCurdy D, Myones BL, Nagy K, Reuman P, Szer I, Travers S, Beutler A, Keenan G, Clark J, Visvanathan S, Fasanmade A, Raychaudhuri A, Mendelsohn A, Martini A, Giannini EH; Paediatric Rheumatology International Trials Organisation; Pediatric Rheumatology Collaborative Study Group. A randomized, placebo-controlled trial of infliximab plus methotrexate for the treatment of polyarticular-course juvenile rheumatoid arthritis. Arthritis Rheum. 2007 Sep;56(9):3096-106. doi: 10.1002/art.22838. PMID 17763439
- [Background] Ruperto N, Lovell DJ, Quartier P, Paz E, Rubio-Perez N, Silva CA, Abud-Mendoza C, Burgos-Vargas R, Gerloni V, Melo-Gomes JA, Saad-Magalhaes C, Sztajnbok F, Goldenstein-Schainberg C, Scheinberg M, Penades IC, Fischbach M, Orozco J, Hashkes PJ, Hom C, Jung L, Lepore L, Oliveira S, Wallace CA, Sigal LH, Block AJ, Covucci A, Martini A, Giannini EH; Paediatric Rheumatology INternational Trials Organization; Pediatric Rheumatology Collaborative Study Group. Abatacept in children with juvenile idiopathic arthritis: a randomised, double-blind, placebo-controlled withdrawal trial. Lancet. 2008 Aug 2;372(9636):383-91. doi: 10.1016/S0140-6736(08)60998-8. Epub 2008 Jul 14. PMID 18632147
- [Background] Lovell DJ, Ruperto N, Goodman S, Reiff A, Jung L, Jarosova K, Nemcova D, Mouy R, Sandborg C, Bohnsack J, Elewaut D, Foeldvari I, Gerloni V, Rovensky J, Minden K, Vehe RK, Weiner LW, Horneff G, Huppertz HI, Olson NY, Medich JR, Carcereri-De-Prati R, McIlraith MJ, Giannini EH, Martini A; Pediatric Rheumatology Collaborative Study Group; Pediatric Rheumatology International Trials Organisation. Adalimumab with or without methotrexate in juvenile rheumatoid arthritis. N Engl J Med. 2008 Aug 21;359(8):810-20. doi: 10.1056/NEJMoa0706290. PMID 18716298
- [Background] Ruperto N, Lovell DJ, Quartier P, Paz E, Rubio-Perez N, Silva CA, Abud-Mendoza C, Burgos-Vargas R, Gerloni V, Melo-Gomes JA, Saad-Magalhaes C, Chavez-Corrales J, Huemer C, Kivitz A, Blanco FJ, Foeldvari I, Hofer M, Horneff G, Huppertz HI, Job-Deslandre C, Loy A, Minden K, Punaro M, Nunez AF, Sigal LH, Block AJ, Nys M, Martini A, Giannini EH; Paediatric Rheumatology International Trials Organization and the Pediatric Rheumatology Collaborative Study Group. Long-term safety and efficacy of abatacept in children with juvenile idiopathic arthritis. Arthritis Rheum. 2010 Jun;62(6):1792-802. doi: 10.1002/art.27431. PMID 20191582
- [Background] Ruperto N, Lovell DJ, Cuttica R, Woo P, Meiorin S, Wouters C, Silverman ED, Balogh Z, Henrickson M, Davidson J, Foeldvari I, Imundo L, Simonini G, Oppermann J, Xu S, Shen YK, Visvanathan S, Fasanmade A, Mendelsohn A, Martini A, Giannini EH; Paediatric Rheumatology INternational Trials Organization (PRINTO); Pediatric Rheumatology Collaborative Study Group (PRCSG). Long-term efficacy and safety of infliximab plus methotrexate for the treatment of polyarticular-course juvenile rheumatoid arthritis: findings from an open-label treatment extension. Ann Rheum Dis. 2010 Apr;69(4):718-22. doi: 10.1136/ard.2009.100354. PMID 20237125
- [Background] Woo P, Southwood TR, Prieur AM, Dore CJ, Grainger J, David J, Ryder C, Hasson N, Hall A, Lemelle I. Randomized, placebo-controlled, crossover trial of low-dose oral methotrexate in children with extended oligoarticular or systemic arthritis. Arthritis Rheum. 2000 Aug;43(8):1849-57. doi: 10.1002/1529-0131(200008)43:83.0.CO;2-F. PMID 10943876
- [Background] Ruperto N, Ravelli A, Castell E, Gerloni V, Haefner R, Malattia C, Kanakoudi-Tsakalidou F, Nielsen S, Bohnsack J, Gibbas D, Rennebohm R, Voygioyka O, Balogh Z, Lepore L, Macejkova E, Wulffraat N, Oliveira S, Russo R, Buoncompagni A, Hilario MO, Alpigiani MG, Passo M, Lovell DJ, Merino R, Martini A, Giannini EH; Pediatric Rheumatology Collaborative Study Group (PRCSG); Paediatric Rheumatology International Trials Organisation (PRINTO). Cyclosporine A in juvenile idiopathic arthritis. Results of the PRCSG/PRINTO phase IV post marketing surveillance study. Clin Exp Rheumatol. 2006 Sep-Oct;24(5):599-605. PMID 17181934
- [Background] Silverman E, Mouy R, Spiegel L, Jung LK, Saurenmann RK, Lahdenne P, Horneff G, Calvo I, Szer IS, Simpson K, Stewart JA, Strand V; Leflunomide in Juvenile Rheumatoid Arthritis (JRA) Investigator Group. Leflunomide or methotrexate for juvenile rheumatoid arthritis. N Engl J Med. 2005 Apr 21;352(16):1655-66. doi: 10.1056/NEJMoa041810. PMID 15843668
- [Background] van Rossum MA, Fiselier TJ, Franssen MJ, Zwinderman AH, ten Cate R, van Suijlekom-Smit LW, van Luijk WH, van Soesbergen RM, Wulffraat NM, Oostveen JC, Kuis W, Dijkstra PF, van Ede CF, Dijkmans BA. Sulfasalazine in the treatment of juvenile chronic arthritis: a randomized, double-blind, placebo-controlled, multicenter study. Dutch Juvenile Chronic Arthritis Study Group. Arthritis Rheum. 1998 May;41(5):808-16. doi: 10.1002/1529-0131(199805)41:53.0.CO;2-T. PMID 9588731
- [Background] Beukelman T, Patkar NM, Saag KG, Tolleson-Rinehart S, Cron RQ, DeWitt EM, Ilowite NT, Kimura Y, Laxer RM, Lovell DJ, Martini A, Rabinovich CE, Ruperto N. 2011 American College of Rheumatology recommendations for the treatment of juvenile idiopathic arthritis: initiation and safety monitoring of therapeutic agents for the treatment of arthritis and systemic features. Arthritis Care Res (Hoboken). 2011 Apr;63(4):465-82. doi: 10.1002/acr.20460. PMID 21452260
- [Background] Giannini EH, Ruperto N, Ravelli A, Lovell DJ, Felson DT, Martini A. Preliminary definition of improvement in juvenile arthritis. Arthritis Rheum. 1997 Jul;40(7):1202-9. doi: 10.1002/1529-0131(199707)40:73.0.CO;2-R. PMID 9214419
- [Background] Wallace CA, Ruperto N, Giannini E; Childhood Arthritis and Rheumatology Research Alliance; Pediatric Rheumatology International Trials Organization; Pediatric Rheumatology Collaborative Study Group. Preliminary criteria for clinical remission for select categories of juvenile idiopathic arthritis. J Rheumatol. 2004 Nov;31(11):2290-4. PMID 15517647
- [Background] Ruperto N, Martini A. Pediatric rheumatology: JIA, treatment and possible risk of malignancies. Nat Rev Rheumatol. 2011 Jan;7(1):6-7. doi: 10.1038/nrrheum.2010.199. Epub 2010 Dec 7. No abstract available. PMID 21135880
- [Background] Diak P, Siegel J, La Grenade L, Choi L, Lemery S, McMahon A. Tumor necrosis factor alpha blockers and malignancy in children: forty-eight cases reported to the Food and Drug Administration. Arthritis Rheum. 2010 Aug;62(8):2517-24. doi: 10.1002/art.27511. PMID 20506368
- [Background] Simard JF, Neovius M, Hagelberg S, Askling J. Juvenile idiopathic arthritis and risk of cancer: a nationwide cohort study. Arthritis Rheum. 2010 Dec;62(12):3776-82. doi: 10.1002/art.27741. PMID 20827782
- [Background] Askling J, Baecklund E, Granath F, Geborek P, Fored M, Backlin C, Bertilsson L, Coster L, Jacobsson LT, Lindblad S, Lysholm J, Rantapaa-Dahlqvist S, Saxne T, van Vollenhoven R, Klareskog L, Feltelius N. Anti-tumour necrosis factor therapy in rheumatoid arthritis and risk of malignant lymphomas: relative risks and time trends in the Swedish Biologics Register. Ann Rheum Dis. 2009 May;68(5):648-53. doi: 10.1136/ard.2007.085852. Epub 2008 May 8. PMID 18467516
- [Background] Askling J, van Vollenhoven RF, Granath F, Raaschou P, Fored CM, Baecklund E, Dackhammar C, Feltelius N, Coster L, Geborek P, Jacobsson LT, Lindblad S, Rantapaa-Dahlqvist S, Saxne T, Klareskog L. Cancer risk in patients with rheumatoid arthritis treated with anti-tumor necrosis factor alpha therapies: does the risk change with the time since start of treatment? Arthritis Rheum. 2009 Nov;60(11):3180-9. doi: 10.1002/art.24941. PMID 19877027
- [Background] Giannini EH, Ilowite NT, Lovell DJ, Wallace CA, Rabinovich CE, Reiff A, Higgins G, Gottlieb B, Singer NG, Chon Y, Lin SL, Baumgartner SW; Pediatric Rheumatology Collaborative Study Group. Long-term safety and effectiveness of etanercept in children with selected categories of juvenile idiopathic arthritis. Arthritis Rheum. 2009 Sep;60(9):2794-804. doi: 10.1002/art.24777. PMID 19714630
- [Derived] Del Giudice E, de Roock S, Vastert SJ, Wulffraat NM, Swart JF, van Dijkhuizen EHP. Patients' and parents' satisfaction to improve patient care in JIA: factors determining acceptable symptom state measured with JAMAR. Rheumatology (Oxford). 2023 May 2;62(5):1920-1925. doi: 10.1093/rheumatology/keac658. PMID 36515484
- [Derived] Giancane G, Papa R, Vastert S, Bagnasco F, Swart JF, Quartier P, Anton J, Kamphuis S, Sanner H, Glerup M, De Benedetti F, Tsitsami E, Remesal A, Moreno E, De Inocencio J, Myrup C, Pallotti C, Kone-Paut I, Franck-Larsson K, Malmstrom H, Cederholm S, Pistorio A, Wulffraat N, Ruperto N; Paediatric Rheumatology International Trials Organisation (PRINTO). Anakinra in Patients With Systemic Juvenile Idiopathic Arthritis: Long-term Safety From the Pharmachild Registry. J Rheumatol. 2022 Apr;49(4):398-407. doi: 10.3899/jrheum.210563. Epub 2022 Feb 1. PMID 35105709
- [Derived] Giancane G, Swart JF, Castagnola E, Groll AH, Horneff G, Huppertz HI, Lovell DJ, Wolfs T, Herlin T, Dolezalova P, Sanner H, Susic G, Sztajnbok F, Maritsi D, Constantin T, Vargova V, Sawhney S, Rygg M, K Oliveira S, Cattalini M, Bovis F, Bagnasco F, Pistorio A, Martini A, Wulffraat N, Ruperto N; Paediatric Rheumatology International Trials Organisation (PRINTO). Opportunistic infections in immunosuppressed patients with juvenile idiopathic arthritis: analysis by the Pharmachild Safety Adjudication Committee. Arthritis Res Ther. 2020 Apr 7;22(1):71. doi: 10.1186/s13075-020-02167-2. PMID 32264969
- [Derived] Swart J, Giancane G, Horneff G, Magnusson B, Hofer M, Alexeeva capital IE, Cyrillic, Panaviene V, Bader-Meunier B, Anton J, Nielsen S, De Benedetti F, Kamphuis S, Stanevica V, Tracahana M, Ailioaie LM, Tsitsami E, Klein A, Minden K, Foeldvari I, Haas JP, Klotsche J, Horne AC, Consolaro A, Bovis F, Bagnasco F, Pistorio A, Martini A, Wulffraat N, Ruperto N; Paediatric Rheumatology International Trials Organisation (PRINTO), BiKeR and the board of the Swedish Registry. Pharmacovigilance in juvenile idiopathic arthritis patients treated with biologic or synthetic drugs: combined data of more than 15,000 patients from Pharmachild and national registries. Arthritis Res Ther. 2018 Dec 27;20(1):285. doi: 10.1186/s13075-018-1780-z. PMID 30587248
- See also: Official website of the Paediatric Rheumatology International Trials Organisation (PRINTO) — http://www.printo.it